CLINICAL TRIAL: NCT00425178
Title: A Phase 1, Open Label, Single Dose, Dose Response, Pilot Study to Evaluate the Safety and Tolerability of Human Fibroblast Growth Factor-1 (FGF-1) in Patients With Diabetic or Venous Stasis Ulcers
Brief Title: FGF-1 for Topical Administration for the Treatment of Diabetic or Venous Stasis Ulcers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CardioVascular BioTherapeutics, Inc. (Industry)
Collaborators: Warren General Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVBT-W2005-01
Record Dates: First submitted 2007-01-18; First posted 2007-01-22 (Estimated); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Chronic Wounds; Diabetes; Venous Stasis Ulcers
Keywords: Chronic wounds; Diabetes; Ulcers; Arterial bypass; Angioplasty; Diabetic ulcers
MeSH Terms: conditions — Diabetes Mellitus; Varicose Ulcer; Ulcer | interventions — Fibroblast Growth Factor 1

INTERVENTIONS:
Drug: FGF-1

SUMMARY:
FGF-1 is being used for the treatment of patients with diabetic or venous stasis ulcers. Procedure includes topical administration of FGF-1 or placebo and evaluation of safety, pharmacokinetics, and wound improvement.

DETAILED DESCRIPTION:
Patients meeting eligibility criteria will be randomized to receive topical administration of either FGF-1 or placebo. Patients will be evaluated at days 1 and 7, post-treatment for safety, pharmacokinetics, and wound healing.

ELIGIBILITY:
Eligibility Criteria:

* Informed consent
* Female patients post-menopausal, sterilized, or on adequate birth control
* Full-thickness lower extremity diabetic or venous statis ulcers of specific target size and of at least 8 weeks but no more than 1 year duration
* Target ulcer freshly debrided at screening or within two weeks prior to screening
* Adequate blood supply defined by transcutaneous oxygen pressure > 20 mmHG and ABI greater than or equal to 0.4
* Compliance with non-weight bearing regimen in diabetic patients
* Compliance with wound care regimen

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-09-02 (Actual); Primary Completion 2006-09-02 (Actual); Study Completion 2006-12-01 (Actual)

PRIMARY OUTCOMES:
Safety
Pharmacokinetics

SECONDARY OUTCOMES:
Wound improvement

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Serena, MD, Principal Investigator — Warren General Hospital
Locations (1):
- Warren General Hospital, Warren, Pennsylvania, United States